CLINICAL TRIAL: NCT04386304
Title: A Phase 1, Open-label, Dose Escalation Study to Evaluate the Safety and Preliminary Efficacy of Orally Administered (+)-Epicatechin in Patients With Becker or Becker-like Muscular Dystrophy With Continued Ambulation Past 16 Years of Age
Brief Title: Safety and Biomarker Response to (+)-Epicatechin in Becker Muscular Dystrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Epirium Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EPM-01-101
Record Dates: First submitted 2020-05-01; First posted 2020-05-13 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Becker Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Catechin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation of (+)-epicatechin (Experimental): Subjects will receive escalating doses of (+)-epicatechin starting at 75 mg/day and progressing to 150 mg/day and 225 mg/day with 2 months treatment duration for each dose. Subjects will continue treatment on the individual's maximum tolerated dose for another 6 months.
  Interventions: Drug: (+)-Epicatechin

INTERVENTIONS:
Drug: (+)-Epicatechin — (+)-Epicatechin is a synthetic flavanol
  Other Names: EB 002; EPM-01

SUMMARY:
This is a Phase 1, open-label, dose escalation study aimed at evaluating the safety, early efficacy and potential biomarkers of (+)-epicatechin in patients with Becker or Becker-like Muscular Dystrophy (BMD).

DETAILED DESCRIPTION:
The safety and tolerability of three escalating doses of (+)-epicatechin will be assessed and early effectiveness measured by changes in plasma biomarkers, tissue biomarkers from muscle biopsies, cardiac imaging, and on clinical function assessments of participants' muscle strength. All patients will receive oral (+)-epicatechin for a total duration of approximately 52 weeks. Three doses of (+)-epicatechin will be tested in sequential 2 month periods with total daily doses of 75, 150, and 225 mg/day (+)-epicatechin. Doses will be escalated every 2 months, if tolerated, for the first 6 months of the study. Participants will then continue to receive the highest does they tolerated for an additional 6 months.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Participant must be ≥16 to <60 years of age.
2. Genotype confirmation showing a mutation of the dystrophin gene.
3. Ambulation - participants must show a history of ambulation past the age of 16 years, with continued ambulation thereafter.
4. If on glucocorticoid treatment in the last 12 months, participants must be on a stable dose at screening. Participants cannot start steroids during the study.

EXCLUSION CRITERIA:

1. A diagnosis of other neurological diseases or presence of relevant somatic disorders that are not related to Becker muscular dystrophy.
2. Participants with a history of migraine headaches requiring medical attention and active treatment within the past 6 months.
3. Participants with allergies to chocolate or cocoa.
4. Surgery or orthopedic injury that might affect muscle strength or function within 3 months before study entry or planned surgery at any time during the study.
5. Presence of a concomitant neurologic disease (e.g., Parkinson's disease) that could negatively impact mobility or balance.
6. Symptomatic heart failure (New York Heart Association Class III or IV) or known left ventricular ejection fraction <40% by echocardiogram.
7. Presence of documented intrinsic lung disease (e.g., chronic obstructive pulmonary disease, pulmonary fibrosis).
8. Evidence of current liver disease or impairment.
9. Inadequate renal function.
10. Platelet count, WBC count, and hemoglobin at Screening <Lower Limit of Normal (LLN).
11. Surgery or orthopedic injury that might affect muscle strength or function within 3 months before study entry or planned surgery at any time during the study

Ages: 16 Years to 59 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Through study completion, up to 1 year
  The TEAEs will be graded using the adult National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

SECONDARY OUTCOMES:
Change in cardiac function as assessed by cardiac magnetic resonance imaging (MRI) | Through study completion, up to 1 year
Change in cardiac function as assessed by plasma biomarkers [e.g. pro-B-type natriuretic peptide (pro-BNP), nitrates]. | Through study completion, up to 1 year
Change in muscle function as assessed by 6-minute walk test (6MWT) | Through study completion, up to 1 year
Change in muscle function as assessed by Time to Run/Walk 10-meter Test (TTRW10) | Through study completion, up to 1 year
Change in muscle function as assessed by Time to 4-stair Climb Test (TT4SC) | Through study completion, up to 1 year
Change in muscle function as assessed by Time to Run/Walk 100-meter Test (TTRW100) | Through study completion, up to 1 year
Change in muscle structure and function as assessed by Western blot analysis of biopsy specimens (e.g. dystrophin expression) | Through study completion, up to 1 year
Change in muscle biomarkers of regeneration in biopsy specimens (e.g. follistatin) | Through study completion, up to 1 year
Change in plasma biomarkers of muscle regeneration (e.g. follistatin, myostatin) | Through study completion, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Epirium Bio Inc.
Locations (3):
- United States (3):
  - UCLA Dept of Human Genetics, Los Angeles, California
  - University of California - Davis Department of Physical Medicine and Rehabilitation, Sacramento, California
  - Washington University School of Medicine, St Louis, Missouri